CLINICAL TRIAL: NCT06792708
Title: A Prospective, Multicenter, Observational Study of LUMRYZ Used in Clinical Practice for the Treatment of Narcolepsy
Brief Title: Observational Study of LUMRYZ in Narcolepsy
Acronym: REFRESH
Status: Active, not recruiting | Type: Observational
Sponsor: Avadel (Industry)
Responsible Party: Sponsor
Other Study IDs: PMLUM-2402
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Starting LUMRYZ: The cohort is comprised of patients prescribed LUMRYZ in clinical practice. All dosing decisions are made by the clinician.
  Interventions: Drug: LUMRYZ

INTERVENTIONS:
Drug: LUMRYZ — Prescribed for narcolepsy in accordance with product label.

SUMMARY:
This is an observational study of LUMRYZ prescribed in clinical practice. Patients are asked if they would be willing to complete questionnaires over a 4-month period after starting LUMRYZ. The questionnaires ask about narcolepsy symptoms, experience with LUMRYZ, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults with narcolepsy
* Oxybate naive or prior treatment with twice-nightly oxybate
* Access to smart phone, tablet or laptop with reliable internet connection
* Able to read/understand English
* Written informed consent and ability to comply with schedule

Exclusion Criteria:

* Already using LUMRYZ
* Clinical or mental health condition excluded by LUMRYZ label
* Any other condition/situation that would adversely impact participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years and older) with a diagnosis of Type 1 or Type 2 narcolepsy
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale | Baseline to Month 4
  Change from the first visit (baseline), prior to start of LUMRYZ, to Month 4; measure of sleepiness with total possible score of 0-24 (higher score equivalent to higher sleepiness)

OTHER OUTCOMES:
Narcolepsy Severity Scale | Baseline to Month 4
  Change from the first visit (baseline), prior to start of LUMRYZ, to Month 4; measure of narcolepsy symptom frequency and impact on daily life with total possible score from 0-57 (higher score indicates more frequent and severe symptoms)
Sheehan Disability Scale | Baseline to Month 4
  Change from the first visit (baseline), prior to start of LUMRYZ, to Month 4; measure of disruption to normal activities using a 0-10 scale, along with the number of days missed and/or underproductive at work/school
Patient Global Impression of Change | Month 4
  Measure of improvement at Month 4 using a scale of 1 (very much improved) to 7 (very much worse); scored by patient
Clinical Global Impression of Change | Month 4
  Measure of improvement at Month 4 using a scale of 1 (very much improved) to 7 (very much worse); scored by clinician
Adverse Reactions | Month 1, Month 2, Month 3, Month 4
  Clinician-directed interview for common adverse reactions

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Jeremy D McConnell, MD PA, Bradenton, Florida
  - Comprehensive Sleep Center, East Lansing, Michigan
  - Patient First MD, Middletown, New Jersey
  - Ghaly Sleep Management Services, East Syracuse, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Abington Neurological Associates, Abington, Pennsylvania
  - Pulmonology Associates, Inc., Wynnewood, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Tricoastal Narcolepsy and Sleep Disorder Center, Sugar Land, Texas
  - Northwest Houston Neurology, Tomball, Texas